CLINICAL TRIAL: NCT06108362
Title: Effect of Intraoperative Terlipressin on the Incidence of Early Postoperative Acute Kidney Injury in Liver Transplantation Patients: a Randomized, Double-blind, Placebo-controlled Study
Brief Title: Effect of Terlipressin on the Incidence of Early Postoperative Acute Kidney Injury in Liver Transplantation Patients
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Beijing Tsinghua Chang Gung Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 23344-4-02
Record Dates: First submitted 2023-10-25; First posted 2023-10-31 (Actual); Last update posted 2023-10-31 (Actual); Status verified 2023-08

CONDITIONS: Acute Kidney Injury; Liver Transplant; Complications
Keywords: terlipressin; Liver Transplant
MeSH Terms: conditions — Acute Kidney Injury | interventions — Terlipressin; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- experimental group (Experimental): Continuous terlipressin infusion，Use a syringe to dilute to 50ml Infusion speed is 2ug/kg*h, From the beginning to the end of the surgery.
  Interventions: Drug: Terlipressin
- control group (Placebo Comparator): Continuous normal saline infusion，Use a syringe to draw 50ml Infusion speed is 4ml/h, From the beginning to the end of the surgery.
  Interventions: Drug: normal saline

INTERVENTIONS:
Drug: Terlipressin — The medication is dispensed by the nursing staff before surgery and given to the anesthesiologist before the procedure begins
  Other Names: Glypressin
  Arms: experimental group
Drug: normal saline — The medication is dispensed by the nursing staff before surgery and given to the anesthesiologist before the procedure begins
  Other Names: normal sodium
  Arms: control group

SUMMARY:
The goal of this clinical trial is to evaluate the effect of intraoperative terlipressin on the incidence of early postoperative acute kidney injury in deceased doner liver transplantation. Patients were randomly divided into experimental group and control group by numerical randomization table. The experimental group was injected with terlipressin perioperative and the control group was injected with placebo

DETAILED DESCRIPTION:
acute kidney injury is a relatively common complication in patients with liver transplantation. Most centers have established prediction models for acute kidney injury after liver transplantation, but the incidence cannot be reduced through perioperative anesthesia management. As an vasopressin receptor agonist, terlipressin can increase blood pressure and improve kidney perfusion at the same time, and perioperative application may reduce the incidence of postoperative acute kidney injury

ELIGIBILITY:
Inclusion Criteria:

* 1) Patients who plan to undergo liver transplantation in our hospital 2) Patients or family members sign informed consent

Exclusion Criteria:

* Patients <18 years old;② Patients undergoing autologous liver transplantation or combined transplantation;③ Patients with lower extremity artery stenosis;(4) Patients with severe heart disease、lung disease、kidney disease;⑤ Patients with severe lung disease;⑥ Patients who used renal replacement therapy before surgery;⑦ the depth of one kidney from the body surface is greater than 4cm;⑧ Patients treated with terlipressin within 2 weeks before surgery⑨ Patients allergic to terlipressin.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 104 (Estimated)
Dates: Start 2023-08-18 (Actual); Primary Completion 2024-06-30 (Estimated); Study Completion 2024-06-30 (Estimated)

PRIMARY OUTCOMES:
Incidence of acute kidney injury after liver transplantation | in 7 days
  acute kidney injury diagnostic criteria (2012 edition)

CONTACTS AND LOCATIONS:
Overall Officials: Huan Zhang, Doctor, Study Chair — department of anesthesia
Locations (1):
- Beijing Tsinghua Chang Gung Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No